CLINICAL TRIAL: NCT05746819
Title: An MRI Ancillary Study of a Malaria Fever Randomized Controlled Trial (RCT)
Brief Title: An MRI Ancillary Study of a Malaria Fever Investigation
Acronym: MRIA
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gretchen Birbeck, Professor, University of Rochester
Other Study IDs: RSRB_STUDY00005384; R01NS111057 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Brain Injuries; Malaria; MRI Imaging; Neurocognitive Deficits; Chronic Kidney Diseases; Behavior Problem
MeSH Terms: conditions — Brain Injuries; Malaria; Renal Insufficiency, Chronic; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Aggressive antipyretics therapy of fever vs usual care in the Malaria RCT study — After clinical trial of the Malaria RCT study, this study will compare children allocated to aggressive antipyretic therapy vs. usual care on the prevalence of structural brain abnormalities after recovery from CNS malaria.
  Other Names: NCT03399318

SUMMARY:
This study will seek consent from parents of children enrolled in the Malaria FEVER study to obtain neuroimaging and 12-month neuropsychiatric outcomes data and kidney function on their child. The imaging and evaluations for this observational study will occur after the child has recovered from the acute malaria infection and has otherwise completed the RCT intervention and safety evaluations.

DETAILED DESCRIPTION:
Despite eradication efforts, ~400,000 African children sustained brain injuries as a result of CNS malaria in 2016. A higher maximum temperature (Tmax) during the acute malaria infection is an established risk factor for neurologic sequelae and a randomized controlled trial (RCT) of aggressive antipyretic therapy with acetaminophen and ibuprofen conducted in Malawi and Zambia began enrollment in 2019 (R01NS102176). In that clinical trial, the primary outcome was Tmax during the acute infection. However, the antipyretic therapies used in this RCT may offer neuroprotective effects without affecting Tmax--for example, neuroprotection through anti-inflammatory mechanisms. In An MRI Ancillary Study of Malaria FEVER RCT, we propose to use neuroimaging in the context of the RCT to further evaluate the potential neuroprotective effects of aggressive antipyretic therapy for CNS malaria and explore possible mechanisms for these effects. Comparing children allocated to aggressive antipyretic therapy vs. usual care on the prevalence of structural brain abnormalities after recovery from CNS malaria will facilitate the evaluation of non-fever pathways for neuroprotection. Brain MRIs will be obtained in children enrolled in the RCT at 1- and 12-months post recovery. Analyses will be completed comparing the odds of having any structural injury based upon RCT treatment allocation and based upon (Tmax) stratified by treatment allocation to assess changes specifically related to response to therapy in terms of fever reduction. Potential mechanisms of aggressive antipyretic-related injury will be evaluated including assessments for treatment-related CNS bleeds. Neuroimaging is a well-established, valid proxy for neurological outcomes after brain injury including in pediatric CNS malaria. Adding this MRI ancillary study to our fever RCT may elucidate mechanisms of treatment-associated injury and allow for early identification of neuroprotection from aggressive antipyretic use that would otherwise require long-term follow-up for cognitive and behavioral assessments. This study will provide critical insights that could inform future neuroprotective studies of malaria that might incorporate imaging to optimize study design. It will also add to our understanding of the long term impact of severe malaria on chronic kidney disease risk in children.

ELIGIBILITY:
Inclusion criteria

1. All children enrolled in the parent Malaria RCT study are eligible
2. Signed parental consent is required
3. CNS symptoms associated with malaria.

Exclusion criteria

1. Circulatory failure (cold extremities, capillary refill > 3 seconds, sunken eyes, ↓ skin turgor)
2. Vomiting in the past 2 hours
3. Serum Cr > 1.2 mg/dL
4. A history of liver disease
5. Jaundice or a total bilirubin of >3.0mg/dL
6. A history of gastric ulcers or gastrointestinal bleeding
7. A history of thrombocytopenia or other primary hematologic disorder
8. Petechiae or other clinical indications of bleeding abnormalities
9. A known allergy to ibuprofen, acetaminophen, aspirin or any non-steroidal medication
10. Any contraindication for nasogastric tube (NGT) placement and/or delivery of enteral medications

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children enrolled in the Malaria RCT who survive to discharge are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
MRI neuroimaging 1a | at 1 month
  Children in the RCT will undergo brain MRIs at 1 month after their acute malaria illness to check for any structural injury following CNS malaria. Two radiologists, blinded to treatment allocation, will independently review images and identify the presence or absence of any injury (present vs absent) For children who are unable to tolerate imaging, brain injury status will be determined by outcomes from age-specific neurocognitive and behavioral assessments.
MRI neuroimaging 1a | at 12 months
  Children in the RCT will undergo brain MRIs at 12 months after their acute malaria illness to check for any structural injury following CNS malaria. Two radiologists, blinded to treatment allocation, will independently review images and identify the presence or absence of any injury (present vs absent) For children who are unable to tolerate imaging, brain injury status will be determined by outcomes from age-specific neurocognitive and behavioral assessments.

SECONDARY OUTCOMES:
Comparing specific abnormalities in the two groups by allocation: Brain atrophy | at 1 month post recovery
  The Potchen volume score is 1-3 abnormal due to atrophy, 4-5 normal, 6-8 edema. And these are analyzed as three ordinal categories--atrophic, normal or edematous
Comparing specific abnormalities in the two groups by allocation: Brain atrophy | at 12 months post recovery
  The Potchen volume score is 1-3 abnormal due to atrophy, 4-5 normal, 6-8 edema. And these are analyzed as three ordinal categories--atrophic, normal or edematous
Comparing specific abnormalities in the two groups by allocation: Gliosis by Fazekas score | 1 month post recovery
  Gliosis by Fazekas score, which assesses white matter lesions on brain MRI scans. The scoring is from 0-3, with 0 = no lesion, 1 = mild, 2 = moderate and 3 = severe.
Comparing specific abnormalities in the two groups by allocation: Gliosis by Fazekas score | 12 month post recovery
  Gliosis by Fazekas score, which assesses white matter lesions on brain MRI scans. The scoring is from 0-3, with 0 = no lesion, 1 = mild, 2 = moderate and 3 = severe.
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in cortical region | at 1 month post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence of regional gliosis or atrophy in cortical region
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in cortical region | at 12 month post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence of regional gliosis or atrophy in cortical region
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in deep gray | 1 month post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence of regional gliosis or atrophy in deep gray
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in deep gray | 12 months post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in deep gray
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in corpus callosum | 1 month post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence of regional gliosis or atrophy in corpus callosum
Comparing specific abnormalities in the two groups by allocation:The presence of or absence regional gliosis or atrophy in corpus callosum | 12 months post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence of regional gliosis or atrophy in corpus callosum
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in posterior fossa | 1 month post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence of regional gliosis or atrophy in posterior fossa
Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in posterior fossa | at 12 months post recovery
  Comparing specific abnormalities in the two groups by allocation:The presence or absence of regional gliosis or atrophy in posterior fossa
Safety assessment: bleeding | at 1-month
  Where GRE imaging is available, we will compare presence/absence of evidence of GRE positive findings
Safety assessment: kidney | At least 6 months post malaria
  Compare incident chronic kidney disease based upon urine albumin:creatinine ratio with a cut off of ACR of 3

CONTACTS AND LOCATIONS:
Overall Officials: Karl B Seydel, PhD, Principal Investigator — Michigan State University, USA
Locations (2):
- Queen Elizabeth Central Hospital, Blantyre, Southern Region, Malawi
- Chipata Central Hospital, Chipata, Eastern Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Research data that documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1-year after study completion
Access Criteria: reasonable written request

REFERENCES:
- [Background] Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York, NY: John Wiley and Sons, 1987.
- [Background] Firth D. Bias reduction of maximum likelihood estimates. Biometrika 1993;80:27-38.
- [Background] Plewes K, Turner GDH, Dondorp AM. Pathophysiology, clinical presentation, and treatment of coma and acute kidney injury complicating falciparum malaria. Curr Opin Infect Dis. 2018 Feb;31(1):69-77. doi: 10.1097/QCO.0000000000000419. PMID 29206655
- [Result] Potchen MJ, Birbeck GL, Demarco JK, Kampondeni SD, Beare N, Molyneux ME, Taylor TE. Neuroimaging findings in children with retinopathy-confirmed cerebral malaria. Eur J Radiol. 2010 Apr;74(1):262-8. doi: 10.1016/j.ejrad.2009.02.010. Epub 2009 Apr 3. PMID 19345538
- [Result] Potchen MJ, Kampondeni SD, Ibrahim K, Bonner J, Seydel KB, Taylor TE, Birbeck GL. NeuroInterp: a method for facilitating neuroimaging research on cerebral malaria. Neurology. 2013 Aug 6;81(6):585-8. doi: 10.1212/WNL.0b013e31829e6ed5. PMID 23918861
- [Result] Birbeck GL, Molyneux ME, Kaplan PW, Seydel KB, Chimalizeni YF, Kawaza K, Taylor TE. Blantyre Malaria Project Epilepsy Study (BMPES) of neurological outcomes in retinopathy-positive paediatric cerebral malaria survivors: a prospective cohort study. Lancet Neurol. 2010 Dec;9(12):1173-1181. doi: 10.1016/S1474-4422(10)70270-2. Epub 2010 Nov 4. PMID 21056005
- [Result] Carter JA, Lees JA, Gona JK, Murira G, Rimba K, Neville BG, Newton CR. Severe falciparum malaria and acquired childhood language disorder. Dev Med Child Neurol. 2006 Jan;48(1):51-7. doi: 10.1017/S0012162206000107. PMID 16359594
- [Result] Carter JA, Mung'ala-Odera V, Neville BG, Murira G, Mturi N, Musumba C, Newton CR. Persistent neurocognitive impairments associated with severe falciparum malaria in Kenyan children. J Neurol Neurosurg Psychiatry. 2005 Apr;76(4):476-81. doi: 10.1136/jnnp.2004.043893. PMID 15774431
- [Result] Carter JA, Neville BG, White S, Ross AJ, Otieno G, Mturi N, Musumba C, Newton CR. Increased prevalence of epilepsy associated with severe falciparum malaria in children. Epilepsia. 2004 Aug;45(8):978-81. doi: 10.1111/j.0013-9580.2004.65103.x. PMID 15270766
- [Result] Dondorp AM, Fanello CI, Hendriksen IC, Gomes E, Seni A, Chhaganlal KD, Bojang K, Olaosebikan R, Anunobi N, Maitland K, Kivaya E, Agbenyega T, Nguah SB, Evans J, Gesase S, Kahabuka C, Mtove G, Nadjm B, Deen J, Mwanga-Amumpaire J, Nansumba M, Karema C, Umulisa N, Uwimana A, Mokuolu OA, Adedoyin OT, Johnson WB, Tshefu AK, Onyamboko MA, Sakulthaew T, Ngum WP, Silamut K, Stepniewska K, Woodrow CJ, Bethell D, Wills B, Oneko M, Peto TE, von Seidlein L, Day NP, White NJ; AQUAMAT group. Artesunate versus quinine in the treatment of severe falciparum malaria in African children (AQUAMAT): an open-label, randomised trial. Lancet. 2010 Nov 13;376(9753):1647-57. doi: 10.1016/S0140-6736(10)61924-1. Epub 2010 Nov 7. PMID 21062666
- [Result] Carter JA, Ross AJ, Neville BG, Obiero E, Katana K, Mung'ala-Odera V, Lees JA, Newton CR. Developmental impairments following severe falciparum malaria in children. Trop Med Int Health. 2005 Jan;10(1):3-10. doi: 10.1111/j.1365-3156.2004.01345.x. PMID 15655008
- [Result] Idro R, Jenkins NE, Newton CR. Pathogenesis, clinical features, and neurological outcome of cerebral malaria. Lancet Neurol. 2005 Dec;4(12):827-40. doi: 10.1016/S1474-4422(05)70247-7. PMID 16297841
- [Result] John CC, Bangirana P, Byarugaba J, Opoka RO, Idro R, Jurek AM, Wu B, Boivin MJ. Cerebral malaria in children is associated with long-term cognitive impairment. Pediatrics. 2008 Jul;122(1):e92-9. doi: 10.1542/peds.2007-3709. Epub 2008 Jun 9. PMID 18541616
- [Result] Severe and complicated malaria. World Health Organization, Division of Control of Tropical Diseases. Trans R Soc Trop Med Hyg. 1990;84 Suppl 2:1-65. No abstract available. PMID 2219249
- [Result] Corbett D, Thornhill J. Temperature modulation (hypothermic and hyperthermic conditions) and its influence on histological and behavioral outcomes following cerebral ischemia. Brain Pathol. 2000 Jan;10(1):145-52. doi: 10.1111/j.1750-3639.2000.tb00251.x. PMID 10668904
- [Result] Greer DM, Funk SE, Reaven NL, Ouzounelli M, Uman GC. Impact of fever on outcome in patients with stroke and neurologic injury: a comprehensive meta-analysis. Stroke. 2008 Nov;39(11):3029-35. doi: 10.1161/STROKEAHA.108.521583. Epub 2008 Aug 21. PMID 18723420
- [Result] Laptook AR, Corbett RJ. The effects of temperature on hypoxic-ischemic brain injury. Clin Perinatol. 2002 Dec;29(4):623-49, vi. doi: 10.1016/s0095-5108(02)00057-x. PMID 12516739
- [Result] Suz P, Vavilala MS, Souter M, Muangman S, Lam AM. Clinical features of fever associated with poor outcome in severe pediatric traumatic brain injury. J Neurosurg Anesthesiol. 2006 Jan;18(1):5-10. doi: 10.1097/01.ana.0000189079.26212.37. PMID 16369134
- [Result] Arrich J, Holzer M, Herkner H, Mullner M. Cochrane corner: hypothermia for neuroprotection in adults after cardiopulmonary resuscitation. Anesth Analg. 2010 Apr 1;110(4):1239. doi: 10.1213/ANE.0b013e3181ce8d34. PMID 20357161
- [Result] Lin ZL, Yu HM, Lin J, Chen SQ, Liang ZQ, Zhang ZY. Mild hypothermia via selective head cooling as neuroprotective therapy in term neonates with perinatal asphyxia: an experience from a single neonatal intensive care unit. J Perinatol. 2006 Mar;26(3):180-4. doi: 10.1038/sj.jp.7211412. PMID 16407967
- [Result] Low E, Boylan GB, Mathieson SR, Murray DM, Korotchikova I, Stevenson NJ, Livingstone V, Rennie JM. Cooling and seizure burden in term neonates: an observational study. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F267-72. doi: 10.1136/archdischild-2011-300716. Epub 2012 Jan 3. PMID 22215799
- [Result] Schulzke SM, Rao S, Patole SK. A systematic review of cooling for neuroprotection in neonates with hypoxic ischemic encephalopathy - are we there yet? BMC Pediatr. 2007 Sep 5;7:30. doi: 10.1186/1471-2431-7-30. PMID 17784966
- [Result] Smit E, Liu X, Jary S, Cowan F, Thoresen M. Cooling neonates who do not fulfil the standard cooling criteria - short- and long-term outcomes. Acta Paediatr. 2015 Feb;104(2):138-45. doi: 10.1111/apa.12784. Epub 2014 Sep 29. PMID 25164710
- [Result] Choi HA, Badjatia N, Mayer SA. Hypothermia for acute brain injury--mechanisms and practical aspects. Nat Rev Neurol. 2012 Feb 28;8(4):214-22. doi: 10.1038/nrneurol.2012.21. PMID 22371279
- [Result] Corry JJ. Use of hypothermia in the intensive care unit. World J Crit Care Med. 2012 Aug 4;1(4):106-22. doi: 10.5492/wjccm.v1.i4.106. eCollection 2012 Aug 4. PMID 24701408
- [Result] Magnusson MO, Dahl ML, Cederberg J, Karlsson MO, Sandstrom R. Pharmacodynamics of carbamazepine-mediated induction of CYP3A4, CYP1A2, and Pgp as assessed by probe substrates midazolam, caffeine, and digoxin. Clin Pharmacol Ther. 2008 Jul;84(1):52-62. doi: 10.1038/sj.clpt.6100431. Epub 2007 Oct 31. PMID 17971810
- [Result] Scaravilli V, Tinchero G, Citerio G; Participants in the International Multi-Disciplinary Consensus Conference on the Critical Care Management of Subarachnoid Hemorrhage. Fever management in SAH. Neurocrit Care. 2011 Sep;15(2):287-94. doi: 10.1007/s12028-011-9588-6. PMID 21755388
- [Result] Chomba E, Haworth A, Atadzhanov M, Mbewe E, Birbeck GL. The socioeconomic status of children with epilepsy in Zambia: implications for long-term health and well-being. Epilepsy Behav. 2008 Nov;13(4):620-3. doi: 10.1016/j.yebeh.2008.06.008. Epub 2008 Aug 12. PMID 18602496
- [Result] Crawley J, Smith S, Kirkham F, Muthinji P, Waruiru C, Marsh K. Seizures and status epilepticus in childhood cerebral malaria. QJM. 1996 Aug;89(8):591-7. doi: 10.1093/qjmed/89.8.591. PMID 8935480
- [Result] Dammann O, Leviton A. Inflammation, brain damage and visual dysfunction in preterm infants. Semin Fetal Neonatal Med. 2006 Oct;11(5):363-8. doi: 10.1016/j.siny.2006.02.003. Epub 2006 Mar 31. PMID 16581321
- [Result] Moxon CA, Chisala NV, Wassmer SC, Taylor TE, Seydel KB, Molyneux ME, Faragher B, Kennedy N, Toh CH, Craig AG, Heyderman RS. Persistent endothelial activation and inflammation after Plasmodium falciparum Infection in Malawian children. J Infect Dis. 2014 Feb 15;209(4):610-5. doi: 10.1093/infdis/jit419. Epub 2013 Sep 17. PMID 24048963
- [Result] Langfitt JT, McDermott MP, Brim R, Mboma S, Potchen MJ, Kampondeni SD, Seydel KB, Semrud-Clikeman M, Taylor TE. Neurodevelopmental Impairments 1 Year After Cerebral Malaria. Pediatrics. 2019 Feb;143(2):e20181026. doi: 10.1542/peds.2018-1026. Epub 2019 Jan 29. PMID 30696757
- [Result] Potchen MJ, Kampondeni SD, Seydel KB, Birbeck GL, Hammond CA, Bradley WG, DeMarco JK, Glover SJ, Ugorji JO, Latourette MT, Siebert JE, Molyneux ME, Taylor TE. Acute brain MRI findings in 120 Malawian children with cerebral malaria: new insights into an ancient disease. AJNR Am J Neuroradiol. 2012 Oct;33(9):1740-6. doi: 10.3174/ajnr.A3035. Epub 2012 Apr 19. PMID 22517285
- [Result] Pongponratn E, Riganti M, Punpoowong B, Aikawa M. Microvascular sequestration of parasitized erythrocytes in human falciparum malaria: a pathological study. Am J Trop Med Hyg. 1991 Feb;44(2):168-75. doi: 10.4269/ajtmh.1991.44.168. PMID 2012260
- [Result] Taylor TE, Fu WJ, Carr RA, Whitten RO, Mueller JS, Fosiko NG, Lewallen S, Liomba NG, Molyneux ME. Differentiating the pathologies of cerebral malaria by postmortem parasite counts. Nat Med. 2004 Feb;10(2):143-5. doi: 10.1038/nm986. Epub 2004 Jan 25. PMID 14745442
- [Result] Medhi N, Das SB, Das RR, Medhi S, Sarma P, Duwara R, Das P, Saikia R. MRI findings of cerebral malaria. A report of two cases. Neuroradiol J. 2009 Aug 29;22(4):407-12. doi: 10.1177/197140090902200408. Epub 2009 Aug 29. PMID 24207146
- [Result] Rasalkar DD, Paunipagar BK, Sanghvi D, Sonawane BD, Loniker P. Magnetic resonance imaging in cerebral malaria: a report of four cases. Br J Radiol. 2011 Apr;84(1000):380-5. doi: 10.1259/bjr/85759874. PMID 21415303
- [Result] Potchen MJ, Kampondeni SD, Seydel KB, Haacke EM, Sinyangwe SS, Mwenechanya M, Glover SJ, Milner DA, Zeli E, Hammond CA, Utriainen D, Lishimpi K, Taylor TE, Birbeck GL. 1.5 Tesla Magnetic Resonance Imaging to Investigate Potential Etiologies of Brain Swelling in Pediatric Cerebral Malaria. Am J Trop Med Hyg. 2018 Feb;98(2):497-504. doi: 10.4269/ajtmh.17-0309. Epub 2018 Jan 4. PMID 29313473
- [Result] Kampondeni SD, Birbeck GL, Seydel KB, Beare NA, Glover SJ, Hammond CA, Chilingulo CA, Taylor TE, Potchen MJ. Noninvasive measures of brain edema predict outcome in pediatric cerebral malaria. Surg Neurol Int. 2018 Mar 1;9:53. doi: 10.4103/sni.sni_297_17. eCollection 2018. PMID 29576904
- [Result] Ibekwe R, Jeaven L, Wilmshurst JM. The role of melatonin to attain electroencephalograms in children in a sub-Saharan African setting. Seizure. 2017 Oct;51:87-94. doi: 10.1016/j.seizure.2017.08.002. Epub 2017 Aug 12. PMID 28826048
- [Result] Gordon SB, Chinula L, Chilima B, Mwapasa V, Dadabhai S, Mlombe Y; Malawi Research Ethics Workshop 2018 Participants. A Malawi guideline for research study participant remuneration. Wellcome Open Res. 2018 Dec 19;3:141. doi: 10.12688/wellcomeopenres.14668.2. eCollection 2018. PMID 30662959
- [Result] Molyneux ME, Taylor TE, Wirima JJ, Borgstein A. Clinical features and prognostic indicators in paediatric cerebral malaria: a study of 131 comatose Malawian children. Q J Med. 1989 May;71(265):441-59. PMID 2690177
- [Result] D'Agostino RB Jr. Propensity score methods for bias reduction in the comparison of a treatment to a non-randomized control group. Stat Med. 1998 Oct 15;17(19):2265-81. doi: 10.1002/(sici)1097-0258(19981015)17:193.0.co;2-b. PMID 9802183
- [Result] Lunceford JK, Davidian M. Stratification and weighting via the propensity score in estimation of causal treatment effects: a comparative study. Stat Med. 2004 Oct 15;23(19):2937-60. doi: 10.1002/sim.1903. PMID 15351954
- [Result] Gladstone M, Lancaster GA, Umar E, Nyirenda M, Kayira E, van den Broek NR, Smyth RL. The Malawi Developmental Assessment Tool (MDAT): the creation, validation, and reliability of a tool to assess child development in rural African settings. PLoS Med. 2010 May 25;7(5):e1000273. doi: 10.1371/journal.pmed.1000273. PMID 20520849
- [Result] Gladstone MJ, Lancaster GA, Jones AP, Maleta K, Mtitimila E, Ashorn P, Smyth RL. Can Western developmental screening tools be modified for use in a rural Malawian setting? Arch Dis Child. 2008 Jan;93(1):23-9. doi: 10.1136/adc.2006.095471. Epub 2007 Mar 22. PMID 17379661
- [Result] Denckla MB. Revised Neurological Examination for Subtle Signs (1985). Psychopharmacol Bull. 1985;21(4):773-800. No abstract available. PMID 4089106
- [Result] Placencia M, Sander JW, Shorvon SD, Ellison RH, Cascante SM. Validation of a screening questionnaire for the detection of epileptic seizures in epidemiological studies. Brain. 1992 Jun;115 ( Pt 3):783-94. doi: 10.1093/brain/115.3.783. PMID 1628202
- [Result] Placencia M, Suarez J, Crespo F, Sander JW, Shorvon SD, Ellison RH, Cascante SM. A large-scale study of epilepsy in Ecuador: methodological aspects. Neuroepidemiology. 1992;11(2):74-84. doi: 10.1159/000110915. PMID 1495577
- [Result] Brim R, Mboma S, Semrud-Clikeman M, Kampondeni S, Magen J, Taylor T, Langfitt J. Cognitive Outcomes and Psychiatric Symptoms of Retinopathy-Positive Cerebral Malaria: Cohort Description and Baseline Results. Am J Trop Med Hyg. 2017 Jul;97(1):225-231. doi: 10.4269/ajtmh.17-0020. PMID 28719298
- [Result] Hosmer DW, Lemeshow, S. Applied Logistical Regression. New York, NY: John Wiley and Sons, 2000.
- [Result] Heinze G, Schemper M. A solution to the problem of separation in logistic regression. Stat Med. 2002 Aug 30;21(16):2409-19. doi: 10.1002/sim.1047. PMID 12210625
- [Result] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Result] Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. Psychol Methods. 2010 Dec;15(4):309-34. doi: 10.1037/a0020761. PMID 20954780
- [Result] MacKinnon DP, Fairchild AJ, Fritz MS. Mediation analysis. Annu Rev Psychol. 2007;58:593-614. doi: 10.1146/annurev.psych.58.110405.085542. PMID 16968208
- [Result] Conroy AL, Opoka RO, Bangirana P, Idro R, Ssenkusu JM, Datta D, Hodges JS, Morgan C, John CC. Acute kidney injury is associated with impaired cognition and chronic kidney disease in a prospective cohort of children with severe malaria. BMC Med. 2019 May 21;17(1):98. doi: 10.1186/s12916-019-1332-7. PMID 31109328
- [Result] Plewes K, Kingston HWF, Ghose A, Wattanakul T, Hassan MMU, Haider MS, Dutta PK, Islam MA, Alam S, Jahangir SM, Zahed ASM, Sattar MA, Chowdhury MAH, Herdman MT, Leopold SJ, Ishioka H, Piera KA, Charunwatthana P, Silamut K, Yeo TW, Lee SJ, Mukaka M, Maude RJ, Turner GDH, Faiz MA, Tarning J, Oates JA, Anstey NM, White NJ, Day NPJ, Hossain MA, Roberts Ii LJ, Dondorp AM. Acetaminophen as a Renoprotective Adjunctive Treatment in Patients With Severe and Moderately Severe Falciparum Malaria: A Randomized, Controlled, Open-Label Trial. Clin Infect Dis. 2018 Sep 14;67(7):991-999. doi: 10.1093/cid/ciy213. PMID 29538635
- [Result] John CC, Park GS, Sam-Agudu N, Opoka RO, Boivin MJ. Elevated serum levels of IL-1ra in children with Plasmodium falciparum malaria are associated with increased severity of disease. Cytokine. 2008 Mar;41(3):204-8. doi: 10.1016/j.cyto.2007.12.008. Epub 2008 Feb 20. PMID 18282763
- [Result] Dobbie M, Crawley J, Waruiru C, Marsh K, Surtees R. Cerebrospinal fluid studies in children with cerebral malaria: an excitotoxic mechanism? Am J Trop Med Hyg. 2000 Feb;62(2):284-90. doi: 10.4269/ajtmh.2000.62.284. PMID 10813486
- [Result] Medana IM, Day NP, Salahifar-Sabet H, Stocker R, Smythe G, Bwanaisa L, Njobvu A, Kayira K, Turner GD, Taylor TE, Hunt NH. Metabolites of the kynurenine pathway of tryptophan metabolism in the cerebrospinal fluid of Malawian children with malaria. J Infect Dis. 2003 Sep 15;188(6):844-9. doi: 10.1086/377583. Epub 2003 Sep 9. PMID 12964115
- [Result] Becker K, Rahlfs S, Nickel C, Schirmer RH. Glutathione--functions and metabolism in the malarial parasite Plasmodium falciparum. Biol Chem. 2003 Apr;384(4):551-66. doi: 10.1515/BC.2003.063. PMID 12751785
- [Result] Greve B, Lehman LG, Lell B, Luckner D, Schmidt-Ott R, Kremsner PG. High oxygen radical production is associated with fast parasite clearance in children with Plasmodium falciparum malaria. J Infect Dis. 1999 Jun;179(6):1584-6. doi: 10.1086/314780. PMID 10228089
- [Result] Clark IA, Mackie EJ, Cowden WB. Injection of free radical generators causes premature onset of tissue damage in malaria-infected mice. J Pathol. 1986 Apr;148(4):301-5. doi: 10.1002/path.1711480406. PMID 3701495
- [Result] Divani AA, Andalib S, Di Napoli M, Lattanzi S, Hussain MS, Biller J, McCullough LD, Azarpazhooh MR, Seletska A, Mayer SA, Torbey M. Coronavirus Disease 2019 and Stroke: Clinical Manifestations and Pathophysiological Insights. J Stroke Cerebrovasc Dis. 2020 Aug;29(8):104941. doi: 10.1016/j.jstrokecerebrovasdis.2020.104941. Epub 2020 May 12. PMID 32689643
- [Result] Gutman JR, Lucchi NW, Cantey PT, Steinhardt LC, Samuels AM, Kamb ML, Kapella BK, McElroy PD, Udhayakumar V, Lindblade KA. Malaria and Parasitic Neglected Tropical Diseases: Potential Syndemics with COVID-19? Am J Trop Med Hyg. 2020 Aug;103(2):572-577. doi: 10.4269/ajtmh.20-0516. Epub 2020 Jun 1. PMID 32484155
- [Result] Seydel KB, Kampondeni SD, Valim C, Potchen MJ, Milner DA, Muwalo FW, Birbeck GL, Bradley WG, Fox LL, Glover SJ, Hammond CA, Heyderman RS, Chilingulo CA, Molyneux ME, Taylor TE. Brain swelling and death in children with cerebral malaria. N Engl J Med. 2015 Mar 19;372(12):1126-37. doi: 10.1056/NEJMoa1400116. PMID 25785970
- [Result] Davids EL, Adams Tucker L, Wambua GN, Fewster DL, Schlebusch L, Karrim SB, Attia M, Nyoni J, Bayouh FG, Kuteesa H, Brahim T, Hoogenhout M, Moussa Kahloul RB, Jearey-Graham N, Gobie HB, Nalugya JS. Child and adolescent mental health in Africa: A qualitative analysis of the perspectives of emerging mental health clinicians and researchers using an online platform. J Child Adolesc Ment Health. 2019 Sep;31(2):93-107. doi: 10.2989/17280583.2019.1659145. PMID 31570090
- [Result] Patel AA, Jannati A, Dhamne SC, Sapuwa M, Kalanga E, Mazumdar M, Birbeck GL, Rotenberg A. EEG markers predictive of epilepsy risk in pediatric cerebral malaria - A feasibility study. Epilepsy Behav. 2020 Dec;113:107536. doi: 10.1016/j.yebeh.2020.107536. Epub 2020 Nov 21. PMID 33232892

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT05746819/Prot_SAP_004.pdf
  • Informed Consent Form: MRI Ancillary Consent Form English Version 4.1 (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT05746819/ICF_001.pdf
  • Informed Consent Form: MRI Ancillary Assent Form English Version 4.0 (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT05746819/ICF_002.pdf